CLINICAL TRIAL: NCT00619333
Title: The Role of Inactive Follicle Stimulating Hormone in Ovarian Dysfunction in Galactosemia
Brief Title: Inactive FSH in Galactosemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Dutch Galactosemia Society (Other)
Responsible Party: Dr. M. E. Rubio-Gozalbo, Academic Hospital Maastricht
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MEC 06-2-073
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Galactosemia; Premature Ovarian Failure
MeSH Terms: conditions — Galactosemias; Primary Ovarian Insufficiency | interventions — Follicle Stimulating Hormone; Luteinizing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: follitropin and lutropin

INTERVENTIONS:
Drug: follitropin and lutropin — follitropin and lutropin

SUMMARY:
The aim of the study is to investigate whether inactive FSH plays a role in the development of Premature Ovarian Failure in women with Classic Galactosemia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of galactosemia through GALT-activity analysis and/or mutation analysis
* Premature Ovarian Failure with FSH > 30 U/l

Exclusion Criteria:

* Gynecological cancers and/or unexplained vaginal bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Estradiol response | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Estela Rubio-Gozalbo, MD, PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Hospital, Maastricht, Netherlands